CLINICAL TRIAL: NCT03301649
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Design, Multiple-Site Clinical Study to Evaluate the Therapeutic Equivalence and Safety of Ivermectin Lotion 0.5% (Actavis Laboratories UT, Inc.) to SKLICE® (Ivermectin) Lotion, 0.5% (Arbor Pharmaceuticals, LLC) in the Treatment of Human Head Lice Infestation
Brief Title: Clinical Endpoint Study of Ivermectin 0.5% Lotion
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Actavis Inc. (Industry)
Collaborators: Teva Pharmaceuticals USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 71691702
Record Dates: First submitted 2017-08-01; First posted 2017-10-04 (Actual); Results first posted 2019-12-20 (Actual); Last update posted 2019-12-20 (Actual); Status verified 2019-12

CONDITIONS: Head Lice
MeSH Terms: interventions — Ivermectin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Generic Ivermectin Lotion 0.5% (Experimental): Infested household participants will administer a single application of up to 117 grams (1 tube) of generic ivermectin 0.5% topical lotion to the dry hair (avoiding contact with eyes) at home on Day 1, leave the lotion on the hair and scalp for 10 minutes, and then rinse off with warm water. Participants will be instructed to wash their hands after application of the study drug, allow hair to dry naturally (pat drying with decontaminated towel is permitted), and to leave hair uncovered after application of the study drug. Following application and rinsing of the study drug, participants are not to shampoo, wash, or rinse their hair or scalp until the Day 2 visit has been completed.
  Interventions: Drug: Generic Ivermectin Lotion 0.5%
- Sklice (Ivermectin) Lotion 0.5% (Active Comparator): Infested household participants will administer a single application of up to 117 grams (1 tube) of Sklice ivermectin 0.5% topical lotion to the dry hair (avoiding contact with eyes) at home on Day 1, leave the lotion on the hair and scalp for 10 minutes, and then rinse off with warm water. Participants will be instructed to wash their hands after application of the study drug, allow hair to dry naturally (pat drying with decontaminated towel is permitted), and to leave hair uncovered after application of the study drug. Following application and rinsing of the study drug, participants are not to shampoo, wash, or rinse their hair or scalp until the Day 2 visit has been completed.
  Interventions: Drug: Sklice® (Ivermectin) Lotion 0.5%
- Vehicle Lotion (Placebo Comparator): Infested household participants will administer a single application of up to 117 grams (1 tube) of vehicle topical lotion to the dry hair (avoiding contact with eyes) at home on Day 1, leave the lotion on the hair and scalp for 10 minutes, and then rinse off with warm water. Participants will be instructed to wash their hands after application of the study drug, allow hair to dry naturally (pat drying with decontaminated towel is permitted), and to leave hair uncovered after application of the study drug. Following application and rinsing of the study drug, participants are not to shampoo, wash, or rinse their hair or scalp until the Day 2 visit has been completed.
  Interventions: Drug: Vehicle Lotion

INTERVENTIONS:
Drug: Generic Ivermectin Lotion 0.5% — Topical lotion, generic formulation of the brand product.
  Arms: Generic Ivermectin Lotion 0.5%
Drug: Sklice® (Ivermectin) Lotion 0.5% — Topical lotion, brand product.
  Arms: Sklice (Ivermectin) Lotion 0.5%
Drug: Vehicle Lotion — Topical lotion, placebo. Has no active ingredient.
  Arms: Vehicle Lotion

SUMMARY:
This clinical study is designed to evaluate the clinical (therapeutic) effect of a generic ivermectin lotion 0.5% (Actavis Laboratories UT, Inc.) relative to that of the Food and Drug Administration (FDA) Reference Listed Drug (RLD) SKLICE® (ivermectin) lotion, 0.5% (Arbor Pharmaceuticals, LLC) in participants with active head lice infestation. Additionally, both the test and reference (that is; the RLD) treatments were tested for superiority to a placebo.

DETAILED DESCRIPTION:
Participants will be randomized by household in a 3:3:1 ratio to receive generic ivermectin lotion 0.5%, Sklice (ivermectin) lotion 0.5%, or vehicle lotion.

ELIGIBILITY:
Inclusion Criteria:

1. Signed Institutional Review Board (IRB)-approved informed consent form that meets all criteria of current FDA regulations. For participants who are considered minors in the state the study is being conducted (<18 years in most states), the parent or legal guardian should sign the consent form and the child will be required to sign a participant "assent" form, as appropriate. Participants 11-17 years of age will read and sign an IRB-approved assent form and participants 6-10 years of age will provide verbal assent. Participants 6 months-5 years of age will be exempt from providing assent based on the child's comprehension and cognitive skills.
2. The participant and/or the participant's parent (legal guardian) is willing to apply the study product as directed, comply with study instructions, and commit to all follow-up visits for the duration of the study.
3. Male or non-pregnant, non-lactating female, 6 months of age or older.
4. Females of childbearing potential must not be pregnant or lactating at Visit 1 (Day -1 to 1) (as confirmed by a negative urine pregnancy test with a sensitivity of less than 50 milli-international units/milliliter [mIU/mL] or equivalent units of human chorionic gonadotropin). Women of childbearing potential must agree to the use of a reliable method of contraception. (for example, total abstinence, intrauterine device, a double-barrier method, oral, transdermal, injected, or implanted non-hormonal or hormonal contraceptive) throughout the study. Female participants using hormonal contraceptives should have been on the same product/dosing regimen for at least 28 days before Visit 1 (Day -1 to 1) and should not change this regimen during the study. A sterile sexual partner is not considered an adequate form of birth control.
5. Index participants (that is, the youngest household member) must have an active head lice infestation, defined as ≥3 live lice (that is, live adults and/or nymphs), at Visit 1 (Day -1 to 1).
6. Household members participating in the study must have ≥1 live louse (that is; live adults and/or nymphs) at Visit 1 (Day -1 to 1).
7. All members of the household must be present for examination. Any male head of household who is unable to attend Visit 1 (Day -1 to 1) may be assessed by a second member of the household as being lice free.

Exclusion Criteria:

1. Females who are pregnant, lactating or planning to become pregnant during the study period.
2. Participants who do not have a known household affiliation with their household members (that is, do not stay in 1 household consistently, sleeping at 1 place several nights and then at another place or location). Household is defined as living in a shared area or space (for example the same house or apartment unit).
3. Any infested member of the household is unable or unwilling to be treated with the study product. This includes male heads of household who do not attend Visit 1 (Day -1 to 1) but report infestation with lice.
4. More than 3 members of the household infested with lice.
5. Presence of visible skin/scalp condition(s) or open wounds at the application site that are not attributable to head lice infestation and that in the opinion of the Investigator will interfere with safety and/or efficacy evaluations.
6. Presence of eczema or atopic dermatitis at the application site.
7. Use of any prescription, over-the-counter, or home remedies for the treatment of head lice within 7 days before Visit 1 (Day -1 to 1).
8. Use of pediculicides within 4 weeks before Visit 1 (Day -1 to 1).
9. Use of systemic anti-parasitic agents within four weeks before Visit 1.
10. Participants with very short (shaved) hair or who are planning to shave head during the study.
11. Use of any hair dye, bleaches, hair straightening, or permanent wave solution on the hair within 14 days before Visit 1 (Day -1 to 1).
12. History of allergy or sensitivity to pediculicides or hair care products.
13. History of any drug hypersensitivity or intolerance that, in the opinion of the Investigator, would compromise the safety of the participant or results of the study.
14. Significant history or current acute or chronic infectious disease, system disorder, Netherton's Syndrome, organ disorder (for example, hepatic or renal impairment) or insufficiency, immunosuppression (from medical treatment or disease), organ transplant, uncontrolled diabetes, uncontrolled hypertension, current ocular condition, or other medical condition that, in the Investigator's opinion, would place the study participant at undue risk by participating in the study.
15. Participants or non-infested household members who would act as the primary caregiver who are of intellectually competent age but unable to understand the protocol requirements, instructions, and study-related restrictions, the nature, scope, and possible consequences of the clinical study.
16. Receipt of any drug as part of a research study within 30 days before Visit 1 (Day -1 to 1).
17. The participant is a member of the investigational study staff or a member of the family of the investigational study staff.
18. Previous participation in this study.

Min Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 905 (Actual)
Dates: Start 2017-10-07 (Actual); Primary Completion 2018-03-12 (Actual); Study Completion 2018-03-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Actavis Inc.
Locations (1):
- Site 1, Miami, Florida, United States

REFERENCES:
- See also: Related Info — https://www.fda.gov/downloads/Drugs/GuidanceComplianceRegulatoryInformation/Guidances/UCM476999.pdf

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 912 infested household participants were included and 911 (905 enrolled [380 index + 525 non-index] + 6 non-enrolled) were treated. Participants were randomized in 3:3:1 to generic ivermectin, Sklice (ivermectin), or vehicle lotion. 1 participant was considered randomized but not dispensed, so not included in any treatment arm.
Pre-assignment Details: Non-enrolled infested participants: Any household member who was infested with lice and agreed to be treated with study drug but did not participate in the study.
  912 infested patients were available to participate in the study, one patient was not dispensed study product, 911 patients (905 enrolled + 6 non-enrolled) were treated.
Groups:
- Generic Ivermectin Lotion 0.5%: Infested household participants administered a single application of up to 117 grams (1 tube) of generic ivermectin 0.5% topical lotion to dry hair (avoiding contact with eyes) at home on Day 1, left the lotion on the hair and scalp for 10 minutes, and then rinsed off with warm water. Participants were instructed to wash their hands after application of the study drug, allow hair to dry naturally (pat drying with decontaminated towel was permitted), and to leave hair uncovered after application of the study drug. Following application and rinsing of the study drug, participants were not to shampoo, wash, or rinse their hair or scalp until the Day 2 visit had been completed.
- Sklice (Ivermectin) Lotion: Infested household participants administered a single application of up to 117 grams (1 tube) of Sklice ivermectin 0.5% topical lotion to dry hair (avoiding contact with eyes) at home on Day 1, left the lotion on the hair and scalp for 10 minutes, and then rinsed off with warm water. Participants were instructed to wash their hands after application of the study drug, allow hair to dry naturally (pat drying with decontaminated towel was permitted), and to leave hair uncovered after application of the study drug. Following application and rinsing of the study drug, participants were not to shampoo, wash, or rinse their hair or scalp until the Day 2 visit had been completed.
- Vehicle Lotion: Infested household participants administered a single application of up to 117 grams (1 tube) of vehicle topical lotion to dry hair (avoiding contact with eyes) at home on Day 1, left the lotion on the hair and scalp for 10 minutes, and then rinsed off with warm water. Participants were instructed to wash their hands after application of the study drug, allow hair to dry naturally (pat drying with decontaminated towel was permitted), and to leave hair uncovered after application of the study drug. Following application and rinsing of the study drug, participants were not to shampoo, wash, or rinse their hair or scalp until the Day 2 visit had been completed.
Period: Overall Study
Arm/Group | Generic Ivermectin Lotion 0.5% | Sklice (Ivermectin) Lotion | Vehicle Lotion
Started | 399 | 400 | 112
Safety Population (Randomized participants who received the study drug.) | 399 | 400 | 112
Modified Intent-to-treat(mITT)Population (Randomized participants, met study criteria, applied study drug, ≥1 post-baseline evaluation visit.) | 372 | 380 | 111
Per-protocol (PP) Population (mITT, made final study visit (Day 15 ± 2 days), and had no significant protocol deviations.) | 345 | 354 | 103
Completed | 356 | 356 | 27
Not Completed | 43 | 44 | 85
Not completed — Need alternate therapy due to live lice | 17 | 25 | 81
Not completed — Lost to Follow-up | 11 | 11 | 3
Not completed — Protocol Violation | 0 | 1 | 1
Not completed — Withdrawal by Subject | 10 | 4 | 0
Not completed — Other than specified | 5 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were randomized and received study drug.
Groups:
- Total: Total of all reporting groups
Arm/Group | Generic Ivermectin Lotion 0.5% | Sklice (Ivermectin) Lotion | Vehicle Lotion | Total
Number analyzed (Participants) | 399 | 400 | 112 | 911
Age, Continuous [Mean (Standard Deviation); unit: years] | 18.8 (15.4) | 16.8 (13.9) | 19.0 (14.4) | 18.2 (14.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 322 | 324 | 97 | 743
  Male | 77 | 76 | 15 | 168
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 344 | 346 | 93 | 783
  Not Hispanic or Latino | 55 | 54 | 19 | 128
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 2
  Asian | 11 | 12 | 3 | 26
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2 | 4
  Black or African American | 6 | 3 | 1 | 10
  White | 377 | 377 | 106 | 860
  More than one race | 3 | 6 | 0 | 9
  Unknown or Not Reported | 0 | 0 | 0 | 0
Number of live lice [Mean (Standard Deviation); unit: live lice] | 4.9 (4.4) | 4.4 (3.5) | 4.5 (3.1) | 4.6 (3.7)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Index Participants Who Were Considered a Treatment Success: PP Population
Description: Treatment success was defined as the absence of live lice. Index participant was defined as the youngest household member who was randomized into the study. Therapeutic equivalence evaluation between test (generic ivermectin lotion 0.5%) and reference groups (Sklice [ivermectin] lotion 0.5%) was done in this endpoint, hence placebo group was not included.
Time Frame: Day 15 ± 2
Population: Index participants in PP population. PP population: randomized participants who met all eligibility criteria, applied study drug, were treatment successes/failures and made the final study visit ( Day 15 ± 2), and had no significant protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Ivermectin Lotion 0.5% | Sklice (Ivermectin) Lotion
Number analyzed (Participants) | 143 | 145
percentage of participants | 90.9 | 89.0
Statistical Analysis 1: Comparison: Generic Ivermectin Lotion 0.5% vs Sklice (Ivermectin) Lotion; If the 90% confidence interval (CI) for the absolute difference between the percentage of participants who were considered a treatment success in the generic ivermectin lotion and sklice (ivermectin) lotion was contained within the range (-20%, +20%) then therapeutic equivalence of the generic ivermectin lotion and sklice (ivermectin) lotion was considered to have been demonstrated; Test type: Equivalence — Therapeutic equivalence was demonstrated if 90% CI of percentage difference between generic ivermectin lotion and sklice (ivermectin) lotion group was within the range (-20%, +20%); Difference in percentage of participants = 1.9, 90% CI 2-sided [-3.9 to 7.8]

2. Primary Outcome: Percentage of Index Participants Who Were Considered a Treatment Success: mITT Population
Description: Treatment success was defined as the absence of live lice. Index participant was defined as the youngest household member who was randomized into the study.
Time Frame: Day 15 ± 2
Population: Index participants in mITT population. mITT population included all randomized participants who met all inclusion/exclusion criteria, applied the study product as instructed, and returned for at least 1 post-baseline evaluation visit.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Ivermectin Lotion 0.5% | Sklice (Ivermectin) Lotion | Vehicle Lotion
Number analyzed (Participants) | 157 | 156 | 49
percentage of participants | 91.7 | 89.7 | 28.6
Statistical Analysis 1: Comparison: Generic Ivermectin Lotion 0.5% vs Vehicle Lotion; Analysis was performed using Cochran- Mantel-Haenszel test, stratified by clinical site in mITT population (using last observation carried forward [LOCF] method); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level
Statistical Analysis 2: Comparison: Sklice (Ivermectin) Lotion vs Vehicle Lotion; Analysis was performed using Cochran- Mantel-Haenszel test, stratified by clinical site in mITT population (using LOCF method); Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level

3. Secondary Outcome: Percentage of All Randomized (Index + Non-Index) Participants Who Were Considered a Treatment Success: PP Population
Description: Treatment success was defined as the absence of live lice. Non-index participant: Any household member who agreed to participate in the study but was not the youngest household member. Index participant: The youngest household member who was randomized into the study. Therapeutic equivalence evaluation between test (generic ivermectin lotion 0.5%) and reference groups (Sklice [ivermectin] lotion 0.5%) was done in this endpoint, hence placebo group was not included.
Time Frame: Day 15 ± 2
Population: PP population: randomized participants who met all eligibility criteria, applied study drug, were treatment successes/failures and made the final study visit (Day 15 ± 2), and had no significant protocol deviations.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Ivermectin Lotion 0.5% | Sklice (Ivermectin) Lotion
Number analyzed (Participants) | 345 | 354
percentage of participants | 91.6 | 90.7
Statistical Analysis 1: Comparison: Generic Ivermectin Lotion 0.5% vs Sklice (Ivermectin) Lotion; If the 90% CI for the absolute difference between the percentage of participants who were considered a treatment success in the generic ivermectin lotion and sklice (ivermectin) lotion was contained within the range (-20%, +20%) then therapeutic equivalence of the generic ivermectin lotion and sklice (ivermectin) lotion was considered to have been demonstrated; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; Difference in percentage of participants = 0.9, 90% CI 2-sided [-2.6 to 4.5]

4. Secondary Outcome: Percentage of All Randomized (Index + Non-Index) Participants Who Were Considered a Treatment Success: mITT Population
Description: Treatment success was defined as the absence of live lice. Non-index participant: Any household member who agreed to participate in the study but was not the youngest household member. Index participant: The youngest household member who was randomized into the study.
Time Frame: Day 15 ± 2
Population: mITT population included all randomized participants who met all inclusion/exclusion criteria, applied the study product as instructed, and returned for at least one post-baseline evaluation visit.
Measure: Number; unit: percentage of participants
Arm/Group | Generic Ivermectin Lotion 0.5% | Sklice (Ivermectin) Lotion | Vehicle Lotion
Number analyzed (Participants) | 372 | 380 | 111
percentage of participants | 92.2 | 91.3 | 25.2
Statistical Analysis 1: Comparison: Generic Ivermectin Lotion 0.5% vs Vehicle Lotion; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level
Statistical Analysis 2: Comparison: Sklice (Ivermectin) Lotion vs Vehicle Lotion; [analysis description as in outcome 2, analysis 2]; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel — Threshold for significance at 0.05 level

ADVERSE EVENTS:
Time Frame: Baseline up to Day 17
Description: Adverse events were collected from participants who were randomized and received the study drug (Safety population).
Arm/Group | Generic Ivermectin Lotion 0.5% | Vehicle Lotion | Sklice (Ivermectin) Lotion
All-Cause Mortality (participants affected / at risk) | 0/399 | 0/400 | 0/112
Serious Adverse Events (participants affected / at risk) | 0/399 | 0/400 | 0/112
Other Adverse Events (participants affected / at risk) | 31/399 | 21/400 | 1/112
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Generic Ivermectin Lotion 0.5% (N=399) | Vehicle Lotion (N=400) | Sklice (Ivermectin) Lotion (N=112)
Eye irritation (Eye disorders) | 2 | 2 | 0
Ocular discomfort (Eye disorders) | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 1 | 0
Vomiting (Gastrointestinal disorders) | 2 | 0 | 0
Application site dysaesthesia (General disorders) | 1 | 2 | 0
Application site erythema (General disorders) | 0 | 1 | 0
Application site exfoliation (General disorders) | 0 | 1 | 0
Application site hypoaesthesia (General disorders) | 0 | 1 | 0
Application site laceration (General disorders) | 1 | 0 | 0
Application site pain (General disorders) | 0 | 1 | 0
Application site paraesthesia (General disorders) | 0 | 1 | 0
Application site pruritus (General disorders) | 9 | 8 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Bacterial infection (Infections and infestations) | 1 | 0 | 0
Ear infection (Infections and infestations) | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 1 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Viral upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0
Headache (Nervous system disorders) | 8 | 2 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study may be published or presented by the Investigator(s) after the review by, and in consultation and agreement with the Sponsor, and such that confidential or proprietary information is not disclosed.

DOCUMENTS (2):
  • Study Protocol (2018-02-01): https://cdn.clinicaltrials.gov/large-docs/49/NCT03301649/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-12): https://cdn.clinicaltrials.gov/large-docs/49/NCT03301649/SAP_001.pdf